CLINICAL TRIAL: NCT00868257
Title: Measurement of Adherence to ART in HIV-Infected School-Aged Children in Uganda
Brief Title: Measurement of Adherence to ART in HIV-Infected Children in Uganda (The CHARTA Study)
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jessica Haberer, MD, Research Scientist/Assistant in Health Decision Sciences, Massachusetts General Hospital
Other Study IDs: R21MH083306 (NIH); R21MH083306 (NIH)
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: HIV; HIV Infections
Keywords: AIDS; Adherence to Antiretroviral Therapy; Pediatric; Resource Limited Setting; Treatment experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples to repeat HIV viral load testing, in the case of processing errors. If these samples are not needed, they may be used for immunologic or viral resistance testing at a future date.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CHARTA study cohort: Primarily 5- to 10-year-old Ugandan children with HIV or AIDS who are taking ART, with some 1- to 4-year-olds included because of recent trends in treating younger children

SUMMARY:
This study will compare methods of determining whether HIV-infected children take their medications.

DETAILED DESCRIPTION:
HIV is a virus that weakens people's immune systems and can cause AIDS. Antiretroviral therapy (ART) is a treatment for HIV that combines different types of antiretroviral medications, but it must be taken throughout a person's life without missing doses to be effective. When people do miss doses, the HIV virus has an opportunity to develop resistance to the medications, making them less effective in the future. Reports indicate that as many as 50% of children infected with HIV who are living in resource-limited countries regularly miss doses of their ART. This study will test different methods for determining children's rates of adherence to ART medications. This will both define the exact magnitude of the problem and direct future efforts in increasing ART adherence in children.

Participation in this study will last 12 months. All children enrolled will undergo a series of assessments of medication adherence. At baseline and every month over the course of the study, researchers will make unannounced home visits to measure the amount of medicine that remains untaken by participants and to record how many times the electronic cap on participants' medication bottles have been removed. Participants with cell phones will also receive monthly phone calls during which they will be asked to measure the amount of their medicine that remains untaken. At study entry and after 6 and 12 months, researchers will also examine child participants' medical records and the results of their regularly scheduled blood tests. At these blood tests, an additional half teaspoon of blood, which may be used in future testing, will be collected and stored by the researchers. After 3, 6, 9, and 12 months, researchers will request to collect hair samples from child participants to test levels of HIV medications in the hair, but participation in this part of the study is optional.

Assessments of reasons for medication adherence will also be performed. At study entry and after 3, 6, 9, and 12 months, children and their parents will complete questionnaires about their understanding of HIV medicines and HIV infection, motivation for the child to take medications, behaviors related to taking medications, and basic personal information. One and 7 months after study entry, some parent participants will also complete interviews with study staff about giving HIV medicines to their children.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Receiving highly active antiretroviral therapy (HAART) through the Children's HIV/AIDS Care Clinic
* Resident in the Mbarara district, defined as living within 30 km or a 2-hour driving radius of the city of Mbarara
* Plans to stay within the Mbarara district for the next year

Exclusion Criteria:

* Attendance at a boarding school

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children recruited from the outpatient Children's HIV/AIDS Care Clinic at the Mbarara University Teaching Hospital in rural, southwestern Uganda
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Median antiretroviral therapy (ART) adherence levels for multiple measures of adherence | Measured monthly for 12 months

SECONDARY OUTCOMES:
Correlation of median ART adherence levels among the multiple measures and with HIV RNA | Measured after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Haberer, MD, MS, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda